CLINICAL TRIAL: NCT05742568
Title: Effects of High-dose Dual Therapy and Bismuth Quadruple Therapy for Helicobacter Pylori Eradication on Intestinal Microecology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20222310-C-1
Record Dates: First submitted 2023-02-03; First posted 2023-02-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Gastritis; Dyspepsia; Helicobacter Pylori Infection; Gastric Cancer; Peptic Ulcer
Keywords: Helicobacter pylori; High-dose dual therapy; Bismuth-combining quadruple therapy; Intestinal Microecology
MeSH Terms: conditions — Gastritis; Dyspepsia; Stomach Neoplasms; Peptic Ulcer | interventions — Esomeprazole; Amoxicillin; Bismuth; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose dual therapy (Experimental): Esomeprazole Enteric Tablets 40mg, 3 times/day; Amoxicillin Capsules 1000mg, 3 times/day.The course of all drugs is two weeks.
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin
- Bismuth Quadruple Therapy (Active Comparator): Esomeprazole Enteric Tablets 40mg, 2 times/day; Amoxicillin Capsules 1000mg, 2 times/day; Clarithromycin Tablets 500mg, 2 times/day; Colloidal Bismuth Tartrate Capsules 220mg, 2 times/day.The course of all drugs is two weeks.
  Interventions: Drug: Bismuth; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Esomeprazole — High-dose dual therapy: given for 14 days at a dose of esomeprazole 20mg 2 tablet TID plus amoxicillin 500 mg 2 capsules TID
  Other Names: Nexium
  Arms: High-dose dual therapy
Drug: Amoxicillin — High-dose dual therapy: given for 14 days at a dose of amoxicillin 500 mg 2 capsules TID plus esomeprazole 20mg 2 tablet TID
  Other Names: Amoxy
  Arms: High-dose dual therapy
Drug: Bismuth — Bismuth-containing quadruple therapy: given for 14 days at a dose of bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 2 tablets BID, amoxicillin 500mg 2 capsules BID and clarithromycin 250mg 2 tablets BID
  Arms: Bismuth Quadruple Therapy
Drug: Esomeprazole — BBismuth-containing quadruple therapy: given for 14 days at a dose of bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 2 tablets BID, amoxicillin 500mg 2 capsules BID and clarithromycin 250mg 2 tablets BID
  Other Names: Nexium
  Arms: Bismuth Quadruple Therapy
Drug: Amoxicillin — Bismuth-containing quadruple therapy: given for 14 days at a dose of bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 2 tablets BID, amoxicillin 500mg 2 capsules BID and clarithromycin 250mg 2 tablets BID
  Arms: Bismuth Quadruple Therapy
Drug: Clarithromycin — Bismuth-containing quadruple therapy: given for 14 days at a dose of bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 2 tablets BID, amoxicillin 500mg 2 capsules BID and clarithromycin 250mg 2 tablets BID
  Arms: Bismuth Quadruple Therapy

SUMMARY:
This study was conducted to investigate the effects of high-dose diphtherapy and bismuth quadruple therapy on H. pylori eradication on intestinal microecology, to clarify the changes in intestinal microbiota diversity and structure before and after the two treatment regimens, and to explore the relationship between different treatment regimens and intestinal microbiota dysbiosis; to further guide the safety and drug resistance of H. pylori eradication by the two treatment regimens. The expected results are to observe the changes of intestinal microbiota diversity and structure before and after treatment with the two treatment regimens.

DETAILED DESCRIPTION:
The trial can be divided into three phases.

1. Enrollment screening phase: patients who had been clearly diagnosed with Hp infection and had not received antibiotic therapy and met the inclusion and exclusion criteria were informed and signed informed consent forms, their basic data information was collected, medical history and laboratory tests before enrollment were taken; if they met the requirements of the trial protocol they were included in the study, and patients' stools were collected for 16S rRNA gene sequencing.
2. Treatment period: Patients were enrolled according to a randomized number table provided in advance by a third party, and patients were randomized in a 1:1 ratio to high-dose diphtherapy and bismuth quadruple therapy to receive 2 weeks of Hp eradication treatment. During the treatment period, patients were provided with written instructions on how to take the medication, instructed on the correct way to take the medication, and improved their compliance; patients were asked to record their symptoms and adverse reactions during the medication period, and were informed of the visiting telephone number and visiting WeChat, so that they could keep in touch with the investigator at any time.
3. Follow-up period: At the end of treatment (i.e., day 14 from the start of treatment), patients were asked to return at that time to have their stools sequenced for 16S rRNA gene, and 6 weeks after the end of treatment (i.e., day 56 from the start of treatment), patients were asked to return at that time to undergo rapid urease test (RUT), 13C/14C-urea breath test (13C/14C-UBT), or fecal Hp antigen test. ) or fecal Hp antigen assay (HpSA), with the results recorded on a CRF form, and the patient's stool collected for 16S rRNA gene sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years, regardless of gender.
2. Patients with definite Hp infection (positive for either 13C/14C urea breath test, rapid urease test, and fecal Hp antigen test) and who have not received H. pylori eradication therapy.
3. Voluntary Hp eradication therapy.
4. Women of childbearing potential are required to use a medically advisable form of contraception during the trial and for 30 days after the trial ends.

Exclusion Criteria:

1. Patients who have had a definite diagnosis of Hp infection and have been treated with antibiotic eradication therapy.
2. Patients with contraindications to or allergies to the study drug.
3. Patients with severe organ damage and complications (e.g., cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine disease
4. Continuous use of anti-ulcer drugs, antibiotics or bismuth complexes (taken at least 2 weeks prior to the screening for Hp infection)
5. Pregnant and lactating women.
6. Having undergone upper gastrointestinal surgery.
7. Have symptoms of dysphagia.
8. Evidence of bleeding or iron deficiency anemia.
9. History of malignancy.
10. History of drug or alcohol abuse within the last 1 year.
11. Systemic application of glucocorticoids, non-steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except for the use of aspirin ≤100 mg/d)
12. Those with psychiatric disorders.
13. Received other clinical trials within the past 3 months
14. Refusal to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in the diversity and structure of fecal microbiota | before treatment,1day after treatment,6 weeks after treatment
  Feces from subjects before treatment , after eradication treatment , and at week 6 after eradication treatment were analyzed for gut microbiota diversity by 16S rRNA gene sequencing, including alpha diversity (representing the abundance of species in the microbial ecosystem, i.e., the number of different species, and evenness, i.e., similar abundance or dominance of some species over others) and beta diversity (representing the difference in microbial composition in one environment compared to another).We will explore the changes in intestinal microbiota diversity and structure before and after treatment with both treatment regimens.

SECONDARY OUTCOMES:
Eradication rate of Helicobacter pylori | 28 days after treatment
  The end point of this study is H.pylori eradication，established by negative [13C] urea breath test （DOB value below 3.9）28 days after the end of eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, Ph. D, Study Director — Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No